CLINICAL TRIAL: NCT06669715
Title: Validation of an Interval Test for Monitoring Cardiovascular Function for Individuals with Different Levels of Physical Fitness
Brief Title: Evaluation of Physical Fitness and Hemodynamics Across a Diverse Population
Acronym: ACT-ON-s1
Status: Recruiting | Type: Observational
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Armin Paravlic, Assistant Professor, PhD, University of Ljubljana
Other Study IDs: ACT-ON; 802-15/2023-5 (Other Grant/Funding Number: University of Ljubljana (slo: Razvojni Sklad UL)); 005-1/2023 (Other: University of Ljubljana (slo: Razvojni Sklad UL))
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Prehypertension (elevated Blood Pressure) or Hypertension; Obesity and Obesity-related Medical Conditions
Keywords: cardiovascular fitness; CRF; physical fitness testing; vascular function; heamodynamics; blood pressure; prehypertension; aerobic capacity; arterial stiffness; endothelial function; post-occlusive reactive hyperemia; PORH
MeSH Terms: conditions — Prehypertension; Hypertension; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asymptomatic individuals - apparently healthy: Asymptomatic individuals - apparently healthy
- Symptomatic individuals: Symptomatic individuals - prehypertensive and hypertensive individuals

SUMMARY:
In this study, investigators will use the IFT 30-15 test, a six-minute walking test, and a treadmill test to assess the participants' cardiorespiratory fitness. For the treadmill cardiopulmonary exercise test (CPET), we will measure indirect gas exchange using a CPET device (K5). Maximum heart rate (HRmax) will be measured with a Polar heart rate monitor (model H10). The six-minute walking test will follow standardized procedures, and the treadmill test will follow a protocol of gradually increasing speed each minute.

The study will involve two groups of participants: healthy individuals and pre-hypertensive individuals. While the IFT 30-15 test has been validated on a diverse range of athletes and physically active individuals, it has not yet been validated in individuals with similar characteristics to our participants (BMI > 30 and limited cardiovascular function). Additionally, a variety of hemodynamic measures and other physical function measures such as sit-to-stand and push-ups will be assessed for all participants.

DETAILED DESCRIPTION:
Study description This study is a work package of the ACT-ON project, aimed at validating different physical fitness assessment tests in diverse populations considering their health status. Thus, in the proposed study we will assess the potential for validating a selected cardiovascular function test for individuals with varying levels of physical fitness. The chosen test, the Intermittent Fitness Test 30-15 (hereafter referred to as IFT 30-15), is a field test commonly used to measure or determine aerobic capacities. More specifically, IFT 30-15 allows for the assessment of maximum oxygen uptake (VO2max), maximum heart rate (HRmax), as well as anaerobic capacity and capacity for intermittent high-intensity running. Of particular importance to us is the test's high potential to determine VO2max and HRmax, which consequently allows for defining workloads in specific training zones.

To collect the necessary data, the investigators will use a range of instruments and tools in all planned studies in the following order:

Upon arrival at the laboratory of the Institute of Sport at the Faculty of Sport, the investigators will measure participants' basic anthropometric characteristics and body composition. the investigators will use a stadiometer and anthropometer (GPM, Model 101, Switzerland) to measure height, and body mass will be measured using a multi-frequency bioelectrical impedance device (InBody 720: Biospace, Korea). Blood pressure will then be measured using the Omron M6 device.

Hemodynamics

Pulse Wave Velocity (PWV) Characteristics

The Vicorder device (software version 4; Skidmore Medical, United Kingdom) will be used to measure pulse wave characteristics (PWA) of the brachial artery and pulse wave velocity from the carotid to the femoral artery (cfPWV). This device uses an oscillometric technique to obtain the pulse wave. cfPWV measurements will be taken using a 10 cm cuff around the upper right thigh to detect the femoral pulse and a 3 cm cuff around the neck to detect the right carotid pulse. The neck cuff is designed to be positioned above one carotid artery, avoiding compression of the trachea and both carotid arteries simultaneously. The distance between the suprasternal notch and the cuff on the upper thigh will be measured according to the manufacturer's instructions. Both cuffs will automatically inflate simultaneously to 65 mmHg, with pulse waves recorded in 3 to 5-second intervals while the participant lies in a supine position.

Flow-Mediated Slowing (FMS)

The VICORDER® EndoCheck FMS model was used for FMS determination. Testing was conducted following the device instructions. The pulse wave velocity (PWV) on the upper arm was measured simultaneously between the wrist and upper part of the right arm over 10 minutes, with a 5-minute flow occlusion period. FMS was determined by continuously measuring the minimal PWV compared to the baseline PWV, with the percentage change designated as FMS.

Physical Performance

Maximal Aerobic Capacity

Equipment for Testing Maximal Aerobic Capacity To obtain physiological parameters, the investigators will use a portable gas analyzer K5 (COSMED, Italy). The device provides reliable values for oxygen uptake (VO2), carbon dioxide production (VCO2), and pulmonary ventilation (VE) on a breath-by-breath basis. Heart rate will simultaneously be measured with a heart rate monitor chest strap (Polar, model H10, Finland). Data will be recorded in 5-second intervals and automatically analyzed using the original Polar software. Similar methods were used in previous studies.

Incremental Treadmill Test

After 5 minutes of baseline measurements while participants stand on the treadmill (HP Cosmos, Germany), participants will warm up at a running speed of 8 km/h and a constant 1% incline. They will then perform the actual test, running to exhaustion while the running speed gradually increases by 2 km/h each minute. VO2peak will be defined as a plateau in VO2 values (decrease < 2.1 ml/kg/min) despite an increase in workload. If this criterion is not met, participants will undergo an additional test at a constant speed equal to or greater than the maximum speed reached at the end of the incremental test, as recommended. Respiratory gases will be continuously measured for each breath during the test and averaged over 10-second intervals. Similar methods were used in previous studies.

30-15 Incremental Fitness Test (30-15IFT)

The 30-15 Incremental Fitness Test (30-15IFT) will be used as a field tool to assess cardiovascular endurance (CRF). This intermittent, incremental test consists of 30-second runs on the spot, followed by 15-second active recovery periods. Running speed will be set at 8 km/h for the first 30-second interval and then increase by 0.5 km/h for each subsequent 30-second interval. Participants will be required to run back and forth between two lines spaced 40 m apart, at a predefined pace determined by a pre-recorded signal. This signal allows participants to adjust their running speed as they enter a 3-meter zone in the middle and at each end of the test field. During the 15-second recovery periods, participants will walk to the nearest line (either in the middle or at the end of the running area, depending on where they finished the previous run), and start the next running phase from this line. Participants will be encouraged to complete as many stages as possible. The test will conclude when the participant can no longer maintain the required running speed or if they fail to reach the 3-meter zone three consecutive times before the beep. The speed of the last successfully completed stage will be recorded as the test result, i.e., the minimal running speed (MRS) during the 30-15IFT (MRS IFT). Similar methods were used in previous studies.

Maximal Aerobic Capacity (VO2max) Using the IFT 30-15 Test

The investigators will measure or determine VO2max indirectly using the following formula:

VO2 max (ml.kg-1.min-1) = 28.3 - (2.15 x S) - (0.741 x L) - (0.0357 x TT) + (0.0586 x L x VIFT) + (1.03 x VIFT) S = gender (male=1, female=2) L = age in years TT = body weight in kilograms VIFT = final speed achieved

6-Minute Walk Test (6MWT)

The protocol for the 6-Minute Walk Test (6MWT) was developed following the American Thoracic Society guidelines (2002). The investigators will check for any contraindications among participants, then ask them to walk as far as they can without running along a 40-meter hallway. If a participant stops walking before the 6 minutes have elapsed (or if the test administrator judges that they should not continue), the reason for stopping will be recorded. Test results will be expressed as the walking distance (i.e., 6MWD) in meters.

Sit-to-stand and Push-ups

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 + years of age) without restriction on sex, health status or physical fitness.

Exclusion Criteria:

* Inability to walk without assistance
* Presence of acute injuries and/or illnesses that limit maximal exertion during physical fitness testing
* Lower extremity injury or surgery within the past 2 years (if not fully rehabilitated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to recruit adults (18 + years of age), without restrictions on sex, health status, or physical fitness level.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity (Vo2max-CPET) | Baseline
  Aerobic capacity will be assessed using cardiopulmonary exercise test on a treadmill. Unit of measure (ml/kg/min)
Aerobic capacity (Vo2max-IFT) | Baseline
  Aerobic capacity will be assessed using 30-15 intermittent fitness test. Unit of measure Vo2max derived from the maximal running velocity at the final stage of the test (ml/kg/min)
Aerobic capacity (Vo2max-6MWT) | Baseline
  Aerobic capacity will be assessed using 6-minute walk test. Unit of measure - Vo2max derived from the maximal walking distance achieved on the text (ml/kg/min)

SECONDARY OUTCOMES:
Stiffness of brachial artery | Baseline
  Brachial artery stiffness measured by pulse wave velocity
Flow-mediated slowing (FMS) of brachial artery | Baseline
  Flow-mediated slowing (FMS) of brachial artery measured by Vicorder device
Brachial artery pulse wave analysis | Baseline
  Brachial artery pulse wave analysis will be assessed using the Vicorder device.
Carotid - femoral (cfPWV) arterial stiffness | Baseline
  cfPWV measured by pulse wave velocity

OTHER OUTCOMES:
Sit-to-stand performance | Baseline
  The sit-to-stand test will be used to assess lower extremity physical performance
Push-ups | Baseline
  Push-ups will be used to assess upper body physical performance

CONTACTS AND LOCATIONS:
Overall Officials: Armin Paravlic, PhD, Principal Investigator — Faculty of Sport, University of Ljubljana
Locations (1):
- Faculty of Sport, University of Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided